CLINICAL TRIAL: NCT03393364
Title: Pain Management in Outpatient Urologic Procedures
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Melody Chen, MD, Urology Resident, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-17-31
Record Dates: First submitted 2017-12-28; First posted 2018-01-08 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Urologic Diseases
MeSH Terms: conditions — Urologic Diseases | interventions — Oxycodone; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid arm (Experimental): Patients receive opioid medication, oxycodone, after outpatient urologic surgery.
  Interventions: Drug: Oxycodone
- Non-opioid arm (Experimental): Patients receive a non-opioid medication, ketorolac, after outpatient urologic surgery.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Oxycodone — Patients receive oxycodone for pain control after outpatient urologic surgery.
  Arms: Opioid arm
Drug: Ketorolac — Patients receive ketorolac for pain control after outpatient urologic surgery
  Arms: Non-opioid arm

SUMMARY:
Goal of this study is to evaluate how pain is controlled after outpatient urologic surgeries. Patients will receive either opioid pain medication or non-opioid medication for pain control. A survey will be conducted at the post-operative appointment to evaluate for pain control.

DETAILED DESCRIPTION:
Patients will be approached in the pre-operative area prior to their outpatient urologic surgery. Informed Consent will be obtained at that time. Patients will be instructed that they will receive a prescription for either opioid pain medication or non-opioid medication for after surgery. The opioid medication includes oxycodone, while the non-opioid includes ketoralac, a non-steroidal anti-inflammatory medication. Subjects will be assigned randomly to either medication. Standard of care after outpatient urologic surgery is either oxycodone or ketoralac, however there is no previous research on whether one is superior than the other. These drugs were chosen because they are the most commonly used medications after outpatient urologic surgery. The study team and patients will not be blinded to the treatment.

They will also receive instructions for non-opioid pain management. If the patients require additional pain medication after surgery, they are instructed to call the provider's office for further evaluation and treatment. The patient's physician will prescribe further medication if warranted. The post-operative appointment is scheduled 2-3 weeks after surgery. At the post-operative appointment, patients will then be given a four question paper survey inquiring how well their pain was managed, how many pills were taken, if any additional non-opioid medications were taken for pain, and how the extra pills were disposed. Other PHI that will be collected includes patient's age, gender, past medical history, past surgical history, renal function, prior medications, and current surgery.

ELIGIBILITY:
Inclusion Criteria:

* outpatient urologic surgery
* age 18 and over

Exclusion Criteria:

* renal dysfunction
* non-English speaking
* employees of organization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Pain control | within 6 weeks of surgery
  Survey evaluating how well pain was controlled

SECONDARY OUTCOMES:
Number of pills used | within 6 weeks of surgery
  Survey evaluating number of pills used

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ponsky, MD, MBA, Study Chair — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided